CLINICAL TRIAL: NCT03907371
Title: The Effect of Donepezil in Radiotherapy-related Cognitive Impairment: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: The Effect of Donepezil in Radiotherapy-related Cognitive Impairment.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019002
Record Dates: First submitted 2019-03-27; First posted 2019-04-09 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Radiation Injuries; Cognitive Impairment
MeSH Terms: conditions — Radiation Injuries; Cognitive Dysfunction | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donepezil (Experimental): Patients receive donepezil with a dosage of 5 milligram at 8 am for one week (Week 1), then 10 milligram at 8 am for 23 weeks (Week 2-24), in the absence of unacceptable toxicity or severe deterioration.
  Interventions: Drug: Donepezil Hydrochloride
- Control (Placebo Comparator): Patients receive placebo with a dosage of one half pill at 8 am for one week (Week 1), then one pill at 8 am for 23 weeks (Week 2-24), in the absence of unacceptable toxicity or severe deterioration.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Donepezil Hydrochloride — Donepezil will be used with a dosage of 5 milligram at 8 am for one week (Week 1), then 10 milligram at 8 am for 23 weeks (Week 2-24).
  Arms: Donepezil
Other: Placebo — Placebo will be used with a dosage of one half pill at 8 am for one week (Week 1), then one pill at 8 am for 23 weeks (Week 2-24).
  Arms: Control

SUMMARY:
Purpose: This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the therapeutic effects of donepezil in radiotherapy-related cognitive impairment.

Further study details as provided by Sun Yat-sen Memorial Hospital, Sun Yat-sen University / Yameitang.

Primary outcome measure: cognitive improvement, which is determined by the difference value of ADAS-cog score before and after the treatment of donepezil.

DETAILED DESCRIPTION:
Application of radiotherapy to patients with head and neck cancer is a mainstay treatment in contemporary oncology practice. However, patients who received radiation are vulnerable to development of cognitive impairment. There is no acknowledged and effective standard treatment for radiotherapy-related cognitive impairment. The investigators supposed that donepezil, as a cholinesterase inhibitor, would relieve radiotherapy-related cognitive impairment after head and neck cancer, and would improve the life quality for these patients and their families.

Primary objectives: This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the efficacy of donepezil on cognition in radiotherapy-related cognitive impairment.

Secondary objectives:

To evaluate the effect of donepezil on sleep disorder, mood disorder, activities of daily living, and safety in patients with radiotherapy-related cognitive impairment.

OUTLINE: This is randomized, double-blind, placebo-controlled clinical trial. Patients will be enrolled and administrated with donepezil or placebo. Donepezil will be supplied as 10 mg per pill to be taken by mouth. Placebo will be supplied as substitute of 10 mg donepezil per pill to be taken by mouth.

Patients will be screened, consented, enrolled and have a washout period for 6 weeks. Then these patients will be randomized to two arms.

Arm І: Patients receive donepezil with a dosage of 5 milligram at 8 am for one week (Week 1), then 10 milligram at 8 am for 23 weeks (Week 2-24), in the absence of unacceptable toxicity or severe deterioration.

Arm ІI: Patients receive placebo with a dosage of one half pill at 8 am for one week (Week 1), then one pill at 8 am for 23 weeks (Week 2-24), in the absence of unacceptable toxicity or severe deterioration.

ELIGIBILITY:
Inclusion Criteria:

* (1) Received radiation therapy due to head and neck cancer.
* (2) Prior irradiation ≥ 1.5 years and ≤ 6 years.
* (3) Age>/= 35 years and age</=60.
* (4) Estimated life expectancy ≥ 12 months.
* (5) Cognitive impairment ≥ 4 weeks, with MMSE total score ≤26, or MoCA total score ≤ 25.
* (6) Routine laboratory studies: normal bilirubin, normal aspartate aminotransferase (AST or SGOT), normal alanine aminotransferase (ALT), normal creatinine, normal white-cell count; normal neutrophils count, normal platelets count; Hb >/=110 gram per millilitres; PT, APTT, INR in a normal range.
* (7) Constant caregivers who well understand and have willingness to sign a written informed consent document.

Exclusion Criteria:

* (1) evidence of tumor metastasis, recurrence, or invasion;
* (2) evidence of very high intracranial pressure that suggests brain hernia and need surgery;
* (3) previous treatment with donepezil or other medications for cognitive impairment;
* (4) history of mental disorders, epilepsy, cognitive impairment before radiotherapy;
* (5) history of stroke, or high risk of vascular dementia;
* (6) family history of Alzheimer's disease, Pick's disease, etc.;
* (7) history of severe head trauma;
* (8) clinically significant active disease, e.g. New York Heart Association Grade II or greater congestive heart failure, serious and inadequately controlled cardiac arrhythmia, bradycardia, significant vascular disease, severe infection;
* (9) history of allergy to relevant drugs;
* (10) pregnancy, lactation, or fertility program in the following 12 months;
* (11) participation in other experimental studies.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 238 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
cognitive change | Baseline to Week 24
  Cognitive change, which is determined by the difference value of ADAS-cog (Alzheimer's Disease Assessment Scale-cognitive subscale) before and after the treatment of donepezil. The rating of ADAS-cog is made on 6-point scale rating from 0 to 5 in 12 domains.

SECONDARY OUTCOMES:
global condition change | Baseline to Week 24
  Efficacy of donepezil on global condition using CIBIC-plus (Clinician's Interview-Based Impression of Change plus). The rating is made on a 7-point scale ranging from "1 = marked improvement" to "7 = marked worsening". A score of "4" indicates no change.
changes of activities of daily living | Baseline to Week 24
  Efficacy of donepezil on activities of daily living using ADL (Activities of Daily Living). Total score is from 0 to 54. The higher score, the lower impairment.
cognition change | Baseline to Week 24
  Efficacy of donepezil on mental statement using MMSE (Mini Mental Status Examination). The total score of MMSE is 30.
psychological statement change | Baseline to Week 24
  Efficacy of donepezil on psychological statement, including sleep disorder, mood disorder etc. using Neuropsychiatric Inventory (NPI) total score.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, M.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided